CLINICAL TRIAL: NCT03046667
Title: Effect of 6 Weeks Daily Consumption of a Cereal-based Juice Beverage on Gastrointestinal Health
Acronym: NEWDRINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Carlsberg Group (Unknown)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M230
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Irritable Bowel
Keywords: Beta glucans; Barley; SCFA; Calprotectin; Microbiota; Hydrogene; Methane; Metabolomics; Stool volume; Stool frequency
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The beverages are provided to the investigator and volunteers with similar color, taste and bottles, only labelled A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drink (Experimental): Test drink: Barley β-glucan
  Interventions: Dietary Supplement: Barley β-glucan
- Control drink (Placebo Comparator): Control drink: barley beverage
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Barley β-glucan — The test beverages with Barley β-glucan is consumed by the participants for the first time at the trial site, followed by a 1 week running-in period were the participants was ingesting half a dose of test drinks. Subsequent were a full dose of the test drinks consumed for 5 weeks. In total was the test drinks consumed for 6 weeks.
  Other Names: barley beta-glucan beverages
  Arms: Test drink
Dietary Supplement: Control — The control beverages is consumed by the participants for the first time at the trial site, followed by a 1 week running-in period were the participants was ingesting half a dose of test drinks. Subsequent were a full dose of the test drinks
  Other Names: barley drink
  Arms: Control drink

SUMMARY:
The project is a randomized, 2-way, blinded parallel trial in which 56 healthy adults of both genders with frequent occurrence of stomach trouble.This intervention trial with 6 weeks of daily intake β-glucans will be carried out with a beverage containing β-glucans and a control beverage without β-glucans. The primary aim is to investigate whether β-glucans from barley has an effect on stomach and intestinal health, including stool volume and frequency. Microbiota, concentrations of short chain fatty acids (butyrate, propionate, acetate), calprotectin, and energy and fat content in feces. Furthermore, blood pressure and exhaled hydrogen and methane, before and after the intervention, subjective perception of gastrointestinal problems and digestion as well as the participants' attitudes towards functional foods are measured using Visual Analog Scale (VAS).

Further, specific metabolites of β-glucans in urine (exploratory endpoint) and certain toxic metabolites from the microbiota using metabolite profiling (metabolomics) are also analyzed

DETAILED DESCRIPTION:
β-glucans from barley slows gastric emptying rate and prolongs the transit time of food in the small intestine." The relatively undigested β-glucans have the ability to increase satiety and stimulate digestion, ensuring regular bowel movements and relieve sluggish bowel movements, including constipation and constipation. β-glucans are fermented down in the large intestine, resulting in production of short-chain fatty acids which inhibit the biosynthesis of cholesterol, hence blood cholesterol levels are lowered (not the goal here). Subsequently, β-glucans may also affect blood pressure. As a direct result of the effects in the intestine, there will be an improvement in the quality of life for people with stomach upsets and maybe a reduction in the risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20 - 27 kg/m2
* Like test and control drink, pasta, meat sauce as these foods are part of the test meal.
* Healthy subjects sometimes or often bothered by mild gastric problems such as bloating, loose stools or constipation
* Willing to handle in 2 x 3-day total feces at the start and end of the study

Exclusion Criteria:

* Suffering from irritable bowel syndrome (IBS), bacterial overgrowth in the small intestine (SIBO) or inflammatory bowel disease (IBD).
* Systemic infections, psychiatric or metabolic diseases, and any clinical condition
* Chronic or frequent use of medication (including blood thinners, excluding contraceptives)
* Frequent loose stools
* Blood donations during or in the month leading up to the study period
* Elite athletes (> 10 hours of hard exercise / week, self-reported)
* High intake of alcohol (defined as a weekly intake of > 7 units for women and > 14 units for men),
* Have or have had a drug addiction
* Participation in other scientific studies during the study period
* Lactating
* Pregnancy or ongoing planning of pregnancy
* Vegetarianism or veganism.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Stool volume | 0 and 6 weeks
  Changes in total stool weight 2 x 3 days from 72 hours before study start and 72 hours before study termination after 6 weeks, determined by a mixed model analysis.

SECONDARY OUTCOMES:
Hydrogen | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min
  Changes in exhaled hydrogen concentrations determined by a mixed model analysis and subsequently at each time point with 0 as a co-variate.
Methane | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min
  Changes in exhaled methane concentrations determined by a mixed model analysis and subsequently at each time point with 0 as a co-variate.
Hydrogen Area Under the Curve | -2, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min
  Area Under the Curve (AUC) for exhaled hydrogen
Methane Area Under the Curve | -2, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min
  Area Under the Curve (AUC) for exhaled methane
Fecal concentrations of SCFA | 0 and 6 weeks
  Changes in SCFA concentrations determined by a mixed model analysis
Determination and variations in fecal microbiota | 0 and 6 weeks
  Changes in microbiota determined by a mixed model analysis
Fecal concentrations of calprotectin | 0 and 6 weeks
  Changes in calprotectin concentrations determined by a mixed model analysis

OTHER OUTCOMES:
Metabolic profile in 24h urine collections | 0 and 6 weeks
  Untargeted metabolic profile of urine samples measured in all samples collected 24 hours before the intervention with beta glucans as well as in samples collected 6 weeks later 24 hours before study termination. The totality of the profiles is used to explore for changes after baseline as detected by multivariate statistics (PLS-DA)
Metabolic profile in 3d fecal collections | 0 and 6 weeks
  Untargeted metabolic profile of fecal samples measured in all samples collected 72-0 hours before the intervention with beta glucans as well as in samples collected 6 weeks later 72-0 hours before study termination. The totality of the profiles is used to explore for changes after baseline as detected by multivariate statistics (PLS-DA)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Ove Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After full anonymization the data may be shared pending acceptance by sponsor approximately 24 months after completion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 24 months from completion
Access Criteria: Full access to published, anonymized data
URL: https://enpadasi.science.ku.dk/